CLINICAL TRIAL: NCT01016405
Title: Cataract and Dry Eye The PHACO Study (Prospective Health Assessment of Cataract Patients' Ocular Surface)
Brief Title: Prospective Health Assessment of Cataract Patients' Ocular Surface
Status: Completed | Type: Observational
Sponsor: Innovative Medical (Industry)
Responsible Party: William Trattler, M.D, The Center for Excellence in Eye Care
Other Study IDs: 0167
Record Dates: First submitted 2009-07-13; First posted 2009-11-19 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Dry Eye
Keywords: Dry eye; incidence and severity; cataract surgery
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Severity of dry eye in patients undergoing cataract surgery

SUMMARY:
This study will determine the incidence and severity of dry eye in patients undergoing cataract surgery as determined by grade on the International Task Force (ITF) scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be at least 55 years old.
* Patients must be scheduled to undergo cataract surgery.

Exclusion Criteria:

* No previous intraocular surgery in the previous 3 months in either eye.
* No previous Corneal laser vision correction in either eye within the last one year.
* No previous lid surgery within the past 3 months.
* Patients may not have used topical antibiotics, topical NSAIDs or topical steroid in either eye in the past month.
* Patients are not eligible if they have recently been started on Restasis solely as a perioperative treatment regimen.
* Patients presently using Restasis in either eye will not undergo any of the study testing but a questionnaire should be completed for these patients regarding use of these medications.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dry eye as evaluated by grade on ITF (International Task Force) level. | One study visit

SECONDARY OUTCOMES:
TBUT (tear break-up time), OSDI (Ocular surface disease index), corneal staining with fluorescein, conjunctival staining with lissamine, Schirmer's, and a patient questionnaire. These are all standard operations of care. | One study visit

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center for Excellence in Eye Care
Locations (1):
- The Center for Excellence in Eye Care, Miami, Florida, United States